CLINICAL TRIAL: NCT05253157
Title: Changes in Pain Interference and Severity After an Episode of Virtual Reality-augmented Remote Rehabilitative Care: a Pragmatic Exploratory Descriptive Trial
Brief Title: Change in Pain With Virtual Reality-augmented Remote Rehabilitative Care
Status: Completed | Type: Observational
Sponsor: XRHealth USA Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: #2022B1014
Record Dates: First submitted 2022-01-21; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-01

CONDITIONS: Musculoskeletal Pain
Keywords: chronic pain; virtual reality; pain management; tele-rehabilitation
MeSH Terms: conditions — Musculoskeletal Pain; Chronic Pain; Agnosia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Virtual Reality Augmented remote rehabilitation — XRHealth offers remote skilled therapy treatments such as education, exercise, and VR-augmented activities. The platform consists of the VRHealth portal with multiple immersive applications for measurement, motor-cognitive training, and mindfulness/cognitive behavioral applications for symptom relief, the external control application, and the XR Health data portal with real-time analytics for evaluating performance. Contraindications for VR use are assessed. Treatment sessions are 60 min long. Duration and frequency are based on clinical judgement. VR interventions used are; VR motor-cognitive: ReAct, Color Match, Memorize, Rotate, and Balloon Blast; VR Reliever: Relax 8, Luna, and Mindset. An external VR portal and mirroring software allows the clinician to view patient activities in real time. Additionally, the clinician can remotely monitor patient performance via the external portal and adjust parameters accordingly.

SUMMARY:
Pain is among the most common chronic conditions in the adult population, often associated with decreased quality of life, functional impairments, increased medication use, increased medical expenditures, and significant economic costs. Due to the worsening opioid crisis, non-pharmacological approaches, such as rehabilitative care, are needed. However, access to in-person rehabilitative care may be limited due to transportation barriers, time constraints, and patient preference to remain at home. The COVID-19 pandemic has further exacerbated barriers to access in-person care, bringing the benefits of tele-rehabilitation into sharper focus. Remote models of care and novel treatment strategies, specifically the utilization of virtual reality (VR) augmented care are emerging as potentially viable treatment alternatives. This paper intends to explore the potential effectiveness of this method of care delivery in patients presenting for rehabilitative care with a primary complaint of pain.

DETAILED DESCRIPTION:
The investigators are proposing a retrospective health and medical records review with a waiver of consent on 52 patients who had remote VR-augmented rehabilitation services from Aug 2020 to Sept of 2021 at XRHealth, a telehealth rehabilitation company utilizing virtual reality applications to augment traditional rehabilitative care. Included patients had an initial and follow-up score on the brief pain interference scale-intensity and severity to explore the association with remote care and changes over time in this validated outcome assessment. In addition, VR headset data will be analyzed to explore the usage and type of VR applications by primary treatment region to help inform the establishment of optimal treatment protocols and explore the association between changes by applications used. De-identified data will be extracted from the proprietary XR Health data portal and will include a unique patient identifier, qualitative and quantitative ratings on the patient experience with XRHealth, number of treatment visits, usage in minutes of the VR applications utilized, and scores on the Brief Pain Inventory: Interference and Severity sub scales. Individual patient records will be reviewed to extract information regarding co-morbidities, condition chronicity, and medications used.

ELIGIBILITY:
Inclusion Criteria:

* presented for treatment at XRHealth with the primary complaint of musculoskeletal pain

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who presented for VR augmented remote rehabilitative care for the primary complaint of musculoskeletal pain.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Brief Pain Inventory: Interference Subscale | Change from baseline in the Brief Pain Inventory: Interference sub scale through study completion, an average of 3 months
  Brief Pain Inventory scale, a self-report scale originally developed to assess pain in individuals with cancer, but has been expanded for assessment of non-
  malignant pain. The subscale of interference assesses how much pain interferes (over the past 24 hrs) with general activity, mood, walking ability, normal work, relations with others, sleep, and enjoyment of life on a scale of: 0=does not interfere up to 10=completely interferes.
Change in Brief Pain Inventory: Severity Subscale | Change from baseline in the Brief Pain Inventory: Severity sub scale through study completion, an average of 3 months
  The severity scale assesses worst, least, average (over the past 24 hours), and current pain on a scale of: 0=no pain up to 10=pain as bad as you can imagine.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna Brown, Principal Investigator — XRHealth USA Inc.
Locations (1):
- XRHealth USA, Inc, Brookline, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yong RJ, Mullins PM, Bhattacharyya N. Prevalence of chronic pain among adults in the United States. Pain. 2022 Feb 1;163(2):e328-e332. doi: 10.1097/j.pain.0000000000002291. PMID 33990113
- [Background] Jette AM. The Role of Nonpharmacological Approaches to Pain Management. Phys Ther. 2018 Nov 1;98(11):907-908. doi: 10.1093/ptj/pzy099. No abstract available. PMID 30321424
- [Background] Lee AC. COVID-19 and the Advancement of Digital Physical Therapist Practice and Telehealth. Phys Ther. 2020 Jul 19;100(7):1054-1057. doi: 10.1093/ptj/pzaa079. No abstract available. PMID 32343836
- [Background] Gumaa M, Rehan Youssef A. Is Virtual Reality Effective in Orthopedic Rehabilitation? A Systematic Review and Meta-Analysis. Phys Ther. 2019 Oct 28;99(10):1304-1325. doi: 10.1093/ptj/pzz093. PMID 31343702
- [Background] Pourmand A, Davis S, Marchak A, Whiteside T, Sikka N. Virtual Reality as a Clinical Tool for Pain Management. Curr Pain Headache Rep. 2018 Jun 15;22(8):53. doi: 10.1007/s11916-018-0708-2. PMID 29904806
- [Background] Keefe FJ, Huling DA, Coggins MJ, Keefe DF, Rosenthal ZM, Herr NR, Hoffman HG. Virtual reality for persistent pain: a new direction for behavioral pain management. Pain. 2012 Nov;153(11):2163-2166. doi: 10.1016/j.pain.2012.05.030. Epub 2012 Jul 4. No abstract available. PMID 22770840
- [Background] Jones T, Moore T, Choo J. The Impact of Virtual Reality on Chronic Pain. PLoS One. 2016 Dec 20;11(12):e0167523. doi: 10.1371/journal.pone.0167523. eCollection 2016. PMID 27997539
- [Background] Garrett B, Taverner T, McDade P. Virtual Reality as an Adjunct Home Therapy in Chronic Pain Management: An Exploratory Study. JMIR Med Inform. 2017 May 11;5(2):e11. doi: 10.2196/medinform.7271. PMID 28495661
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Tan G, Jensen MP, Thornby JI, Shanti BF. Validation of the Brief Pain Inventory for chronic nonmalignant pain. J Pain. 2004 Mar;5(2):133-7. doi: 10.1016/j.jpain.2003.12.005. PMID 15042521
- [Background] Keller S, Bann CM, Dodd SL, Schein J, Mendoza TR, Cleeland CS. Validity of the brief pain inventory for use in documenting the outcomes of patients with noncancer pain. Clin J Pain. 2004 Sep-Oct;20(5):309-18. doi: 10.1097/00002508-200409000-00005. PMID 15322437
- [Background] Jaeschke R, Singer J, Guyatt GH. Measurement of health status. Ascertaining the minimal clinically important difference. Control Clin Trials. 1989 Dec;10(4):407-15. doi: 10.1016/0197-2456(89)90005-6. PMID 2691207